CLINICAL TRIAL: NCT02482909
Title: A Prospective Randomized Study to Compare the Efficacy of Radiofrequency Ablation and Hepatic Resection as a Primary Treatment for Single Small Hepatocellular Carcinoma
Brief Title: A Study Comparing Radiofrequency Ablation and Hepatic Resection for Hepatocellular Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The post-treatment recurrence rate was expected to be different between two treatment groups.
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Kyung-Suk Suh, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0520090
Record Dates: First submitted 2015-06-20; First posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hepatic resection (Experimental): Hepatic resection is performed as a primary treatment for hepatocellular carcinoma.
  Interventions: Procedure: Hepatic resection
- Radiofrequency ablation (Experimental): Radiofrequency ablation is performed as a primary treatment for hepatocellular carcinoma.
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Hepatic resection — Anatomical surgical resection of the liver including the tumor
  Arms: Hepatic resection
Procedure: Radiofrequency ablation — Percutaneous ablation using radiofrequency under the imaging guidance
  Arms: Radiofrequency ablation

SUMMARY:
The purpose of this prospective randomized study is to compare the efficacy and safety of radiofrequency ablation and hepatic resection for small hepatocellular carcinomas with very homogeneous underlying conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 70 years
2. Child-Pugh class A (score 5-6)
3. Single hepatocellular carcinoma
4. Maximal diameter of the tumor from 2 to 4 cm when measured on MRI or CT (The diameter on MRI was measured prior to that on CT)
5. No previous treatment
6. Platelet count > 80,000/mm3

Exclusion Criteria:

1. HCC abutting main hepatic veins or the first branches of the main portal vein
2. HCC abutting vessels ≥ 0.5 cm

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2005-07; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The patient survival | From the intervention up to 5 years or until the death of the participant whichever came first

SECONDARY OUTCOMES:
The disease-free survival | From the intervention up to 5 years or until hepatocellular carcinoma recurrence whichever came first

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Suk Suh, ME, PhD, Study Director — Seoul National University Hospital